CLINICAL TRIAL: NCT00929864
Title: A Randomized, Head-to-Head, Single-Blind Study to Compare the Efficacy and Safety of Subcutaneous Abatacept Versus Subcutaneous Adalimumab, Both With Background Methotrexate, in Biologic-Naive Subjects With Rheumatoid Arthritis
Brief Title: Abatacept Versus Adalimumab Head-to-Head
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IM101-235
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Results first posted 2014-01-03 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Adalimumab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abatacept (Active Comparator)
  Interventions: Drug: Abatacept
- Adalimumab (Active Comparator)
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Abatacept — Syringes, Subcutaneous, 125 mg/syringe for Subcutaneous, Weekly Subcutaneous injections, 24 months (729 days)
  Other Names: Orencia; BMS-188667
  Arms: Abatacept
Drug: Adalimumab — Syringes, Subcutaneous, 40 mg, Biweekly Subcutaneous injections, 24 months (729 days)
  Other Names: Humira
  Arms: Adalimumab

SUMMARY:
The purpose of this study is demonstrate that subcutaneous abatacept is non-inferior (no worse than) to subcutaneous adalimumab in the treatment of subjects with rheumatoid arthritis who are biologic naive

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe Rheumatoid arthritis (RA) according to American College of Rheumatology (ACR) criteria
* Methotrexate failure
* Naive to RA biologics
* ≤5 years duration of disease
* Disease Activity Score-28 C-reactive protein (DAS28 CRP) ≥ 3.2
* Willingness to self-inject subcutaneous (SC) drug

Exclusion Criteria:

* Previous or current medical conditions that are warnings against the use of tumor necrosis factor (TNF)-blocking agents
* History of active or chronic hepatitis
* Cancer in the last 5 years
* History of severe chronic or recurrent bacterial or viral infections
* Risk of tuberculosis
* Current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, Gastro-intestinal, pulmonary, cardiac, neurologic, or cerebral disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 869 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (80):
- United States (63):
  - Rheumatology Associates, Pc, Birmingham, Alabama
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Clinical And Translational Research Center Of Alabama, Pc, Tuscaloosa, Alabama
  - Sun Valley Arthritis Center, Ltd., Peoria, Arizona
  - Mercy Clinic Hot Springs Communities, Hot Springs, Arkansas
  - Talbert Medical Group, Huntington Beach, California
  - Allergy & Rheumatology Medical Clinic, Inc., La Jolla, California
  - Valerius Med Group & Res Ctr Of Greater Long Beach, Inc., Long Beach, California
  - Irene Y. Tong, Pasadena, California
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Healthcare Partners Medical Group, Torrance, California
  - Drs. Goldin, Nies, Klashman & Eng, Torrance, California
  - Inland Rheumatology & Osteoporosis Medical Group, Upland, California
  - Arthritis And Rheumatic Disease Specialties, Aventura, Florida
  - University Of Florida College Of Medicine At Jacksonville, Gainesville, Florida
  - Center For Arthritis And Rheumatic Diseases, Miami, Florida
  - Arthritis Research Of Florida, Inc., Palm Harbor, Florida
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Miami Research Associates, South Miami, Florida
  - West Broward Rheumatology Associates, Tamarac, Florida
  - Lovelace Scientific Resources, Inc, Venice, Florida
  - Arthritis & Rheumatology Of Georgia, Atlanta, Georgia
  - Laureate Clinical Research Group, Atlanta, Georgia
  - Arthritis Center Of North Georgia, Gainesville, Georgia
  - St. Luke'S Clinic - Rheumatology, Boise, Idaho
  - Coeur D'Alene Arthrit Clin, Coeur d'Alene, Idaho
  - Quincy Medical Group, Quincy, Illinois
  - Rockford Orthopedic Associates, Ltd., Rockford, Illinois
  - Physicians Clinic Of Iowa, Cedar Rapids, Iowa
  - Center For Arthritis And Osteoporosis, Elizabethtown, Kentucky
  - Bluegrass Community Research, Inc., Lexington, Kentucky
  - Klein And Associates, M.D., Pa, Cumberland, Maryland
  - The Center For Rheumatology And Bone Research, Wheaton, Maryland
  - Brigham And Women'S Hospital, Boston, Massachusetts
  - Mansfield Health Center, Mansfield, Massachusetts
  - Associated Internal Medicine Specialists, Battle Creek, Michigan
  - Rheumatology Pc, Kalamazoo, Michigan
  - Arthritis Associates Of Mississippi, Jackson, Mississippi
  - Physician Groups, Lc Dba, St Louis, Missouri
  - Arthritis Center Of Reno, Reno, Nevada
  - Seacoast Arthritis And Osteoporosis Center, Dover, New Hampshire
  - Nashua Rheumatology, Nashua, New Hampshire
  - Arthritis And Osteoporosis Associates Of New Mexico, Las Cruces, New Mexico
  - North Shore Lij Health System, Lake Success, New York
  - Winthrop University Hospital, Mineola, New York
  - Rheumatology Associates Of Long Island, Smithtown, New York
  - Asheville Rheumatology & Osteoporosis Research Asso P. A., Asheville, North Carolina
  - Carolina Pharmaceutical Research, Statesville, North Carolina
  - Health Research Of Oklahoma, Oklahoma City, Oklahoma
  - Health Research Institute, Oklahoma City, Oklahoma
  - Lynn Health Sciences Institute, Oklahoma City, Oklahoma
  - East Penn Rheumatology Associates, P.C., Bethlehem, Pennsylvania
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center Of Reading, Llp, Wyomissing, Pennsylvania
  - Low Country Rheumatology, Pa, Charleston, South Carolina
  - Columbia Arthritis Center, P.A., Columbia, South Carolina
  - Lovelace Scientific Resources, Inc., Austin, Texas
  - Arthritis Centers Of Texas, Dallas, Texas
  - Rheumatic Disease Clinical Research Center, Llc, Houston, Texas
  - Center For Arthritis & Rheumatic Diseases, Pc, Chesapeake, Virginia
  - Rockwood Research Center, Spokane, Washington
  - Mountain State Clinical Research, Clarksburg, West Virginia
  - Rheumatic Disease Center, Glendale, Wisconsin
- Argentina (9):
  - Local Institution, Ciudad Autonoma de Beunos Aire, Buenos Aires
  - Local Institution, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Local Institution, Ciudad Autonoma, Buenos Aires
  - Local Institution, Quilmes, Buenos Aires
  - Local Institution, Cordoba, Crd, Córdoba Province
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, San Juan, San Juan Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, San Miguel de Tucumán, Tucumán Province
- Canada (4):
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Hamilton, Ontario
  - Local Institution, Québec, Quebec
  - Local Institution, Trois-Rivières, Quebec
- Local Institution, Santiago, Providencia, Chile
- Peru (3):
  - Local Institution, Bellavista, Callao 2
  - Local Institution, Lima, Lima Province
  - Local Institution, Lima

REFERENCES:
- [Derived] Jabado O, Maldonado MA, Schiff M, Weinblatt ME, Fleischmann R, Robinson WH, He A, Patel V, Greenfield A, Saini J, Galbraith D, Connolly SE. Differential Changes in ACPA Fine Specificity and Gene Expression in a Randomized Trial of Abatacept and Adalimumab in Rheumatoid Arthritis. Rheumatol Ther. 2022 Apr;9(2):391-409. doi: 10.1007/s40744-021-00404-x. Epub 2021 Dec 8. PMID 34878629
- [Derived] Keystone EC, Ahmad HA, Yazici Y, Bergman MJ. Disease activity measures at baseline predict structural damage progression: data from the randomized, controlled AMPLE and AVERT trials. Rheumatology (Oxford). 2020 Aug 1;59(8):2090-2098. doi: 10.1093/rheumatology/kez455. PMID 31819995
- [Derived] Fleischmann R, Weinblatt M, Ahmad H, Maldonado MA, Alemao E, Ye J, Schiff M. Efficacy of Abatacept and Adalimumab in Patients with Early Rheumatoid Arthritis With Multiple Poor Prognostic Factors: Post Hoc Analysis of a Randomized Controlled Clinical Trial (AMPLE). Rheumatol Ther. 2019 Dec;6(4):559-571. doi: 10.1007/s40744-019-00174-7. Epub 2019 Oct 22. PMID 31642045
- [Derived] Fleischmann R, Connolly SE, Maldonado MA, Schiff M. Brief Report: Estimating Disease Activity Using Multi-Biomarker Disease Activity Scores in Rheumatoid Arthritis Patients Treated With Abatacept or Adalimumab. Arthritis Rheumatol. 2016 Sep;68(9):2083-9. doi: 10.1002/art.39714. PMID 27111089
- [Derived] Schiff M, Weinblatt ME, Valente R, Citera G, Maldonado M, Massarotti E, Yazici Y, Fleischmann R. Reductions in disease activity in the AMPLE trial: clinical response by baseline disease duration. RMD Open. 2016 Apr 19;2(1):e000210. doi: 10.1136/rmdopen-2015-000210. eCollection 2016. PMID 27110385
- [Derived] Fleischmann R, Weinblatt ME, Schiff M, Khanna D, Maldonado MA, Nadkarni A, Furst DE. Patient-Reported Outcomes From a Two-Year Head-to-Head Comparison of Subcutaneous Abatacept and Adalimumab for Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2016 Jul;68(7):907-13. doi: 10.1002/acr.22763. PMID 26473625
- [Derived] Sokolove J, Schiff M, Fleischmann R, Weinblatt ME, Connolly SE, Johnsen A, Zhu J, Maldonado MA, Patel S, Robinson WH. Impact of baseline anti-cyclic citrullinated peptide-2 antibody concentration on efficacy outcomes following treatment with subcutaneous abatacept or adalimumab: 2-year results from the AMPLE trial. Ann Rheum Dis. 2016 Apr;75(4):709-14. doi: 10.1136/annrheumdis-2015-207942. Epub 2015 Sep 10. PMID 26359449
- [Derived] Schiff M, Weinblatt ME, Valente R, van der Heijde D, Citera G, Elegbe A, Maldonado M, Fleischmann R. Head-to-head comparison of subcutaneous abatacept versus adalimumab for rheumatoid arthritis: two-year efficacy and safety findings from AMPLE trial. Ann Rheum Dis. 2014 Jan;73(1):86-94. doi: 10.1136/annrheumdis-2013-203843. Epub 2013 Aug 20. PMID 23962455
- [Derived] Weinblatt ME, Schiff M, Valente R, van der Heijde D, Citera G, Zhao C, Maldonado M, Fleischmann R. Head-to-head comparison of subcutaneous abatacept versus adalimumab for rheumatoid arthritis: findings of a phase IIIb, multinational, prospective, randomized study. Arthritis Rheum. 2013 Jan;65(1):28-38. doi: 10.1002/art.37711. PMID 23169319
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 28-October-2009 to 23-November-2012. Study conducted in biologic-naive participants with Rheumatoid Arthritis (RA) who have failed on methotrexate therapy.
Pre-assignment Details: 869 enrolled; 648 randomized; 646 randomized and treated. Reasons for not randomized: 4 pregnancy; 23 lost to follow-up; 133 administrative reasons by Sponsor; 4 no longer met study criteria; 7 other; 50 had reasons missing. Two participants randomized/not treated: no longer met study criteria. Randomization stratified by DAS28-CRP>5.1, <=5.1
Groups:
- 125 mg Abatacept SC Weekly: Abatacept 125 mg weekly subcutaneous (SC) self administered injections for 24 months (729 days). Methotrexate (MTX) was co-administered; a stable dose of maximum tolerated methotrexate (minimum of 15 mg and maximum of 25 mg) per week. Participants were allowed to enroll with MTX doses <15 mg/week but >= 7.5 mg/week if intolerance to higher doses was documented. Participants could also enroll while receiving hydrochloroquine or sulfasalazine in addition to MTX.
- 40 mg Adalimumab SC Biweekly: Adalimumab 40 mg, biweekly (every 14 days) subcutaneous (SC) self administered injections for 24 months (729 days). Methotrexate (MTX) was co-administered; a stable dose of maximum tolerated methotrexate (minimum of 15 mg and maximum of 25 mg) per week. Participants were allowed to enroll with MTX doses <15 mg/week but >= 7.5 mg/week if intolerance to higher doses was documented. Participants could also enroll while receiving hydrochloroquine or sulfasalazine in addition to MTX.
Period: Overall Study
Arm/Group | 125 mg Abatacept SC Weekly | 40 mg Adalimumab SC Biweekly
Started | 318 | 328
Completed | 252 | 245
Not Completed | 66 | 83
Not completed — Death | 1 | 1
Not completed — Adverse Event | 11 | 30
Not completed — Lack of Efficacy | 19 | 16
Not completed — Lost to Follow-up | 7 | 12
Not completed — Withdrawal by Subject | 20 | 9
Not completed — No longer met criteria | 2 | 1
Not completed — Poor or non-compliance | 3 | 3
Not completed — Pregnancy | 0 | 3
Not completed — Administrative reason by Sponsor | 1 | 1
Not completed — Non-specified | 2 | 7

BASELINE CHARACTERISTICS:
Population: All randomized and treated participants who started the 12 month period.
Groups:
- Abatacept: Abatacept 125 mg weekly subcutaneous (SC) self administered injections for 24 months (729 days). Methotrexate (MTX) was co-administered; a stable dose of maximum tolerated methotrexate (minimum of 15 mg and maximum of 25 mg) per week. Participants were allowed to enroll with MTX doses <15 mg/week but >= 7.5 mg/week if intolerance to higher doses was documented. Participants could also enroll while receiving hydrochloroquine or sulfasalazine in addition to MTX.
- Adalimumab: Adalimumab 40 mg, bi-weekly (every 14 days) subcutaneous (SC) self administered injections for 24 months (729 days). Methotrexate (MTX) was co-administered; a stable dose of maximum tolerated methotrexate (minimum of 15 mg and maximum of 25 mg) per week. Participants were allowed to enroll with MTX doses <15 mg/week but >= 7.5 mg/week if intolerance to higher doses was documented. Participants could also enroll while receiving hydrochloroquine or sulfasalazine in addition to MTX.
- Total: Total of all reporting groups
Arm/Group | Abatacept | Adalimumab | Total
Number analyzed (Participants) | 318 | 328 | 646
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (12.6) [19 to 83] | 51.0 (12.8) [19 to 85] | 51.2 (12.7) [19 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 270 | 529
  Male | 59 | 58 | 117
Region of Enrollment [Number; unit: participants]
  North America | 230 | 235 | 465
  South America | 88 | 93 | 181

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants Meeting the American College of Rheumatology (ACR) Criteria of 20% Improvement (ACR20) After 12 Months of Treatment - Intent to Treat Population
Description: Proportion(%)=number of participants meeting criteria (n) divided by number of participants who received drug (N). The ACR score indicates degree of improvement in a patient's rheumatoid arthritis (RA), based on guidelines set forth by the ACR and represents a percentage. To qualify a ACR20 score, patient must have >=20% fewer tender joints and >=20% fewer swollen joints and show 20% improvement from baseline in at least 3 of: patient overall assessment of his/her RA, physician global assessment of the patient's RA, patient self-assessment of pain, patient self-assessment of physical functioning, and results of an erythrocyte sedimentation rate or C-reactive protein (CRP) test (to assess inflammation). Baseline was Day 1. Randomization was stratified using screening Disease Activity Score-28 (DAS28) CRP, a composite of 4 variables: number of tender joints/28, number of swollen joints/28, CRP in mg/L and participant assessment of disease activity with visual analogue scale.
Time Frame: Day 1 to Day 365
Population: The intent to treat (ITT) analysis population was defined as all participants randomized into the study who received at least one dose of study drug. n/N = 206/318 and 208/328 in the abatacept and adalimumab arms, respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abatacept | Adalimumab
Number analyzed (Participants) | 318 | 328
percentage of participants | 64.8 [59.5 to 70.0] | 63.4 [58.2 to 68.6]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab; The null and alternative hypotheses are H0: T - C<= δ vs. Ha:T - C > δ, where T is the treatment effect of abatacept, C is the effect of active control (adalimumab),and δ is non-inferiority margin. Abatacept is defined as δ non-inferior to adalimumab when H0 is rejected. More specifically, if the lower bound of the 95% two-sided confidence interval for C-T is greater than δ,, then that Abatacept is δ non-inferior to adalimumab can be claimed; Test type: Non-Inferiority or Equivalence — Analysis tested for non-inferiority. Abatacept will be considered non-inferior to adalimumab if the upper limit of the 95% two-sided CI of difference in ACR20 response rates between the adalimumab arm and the abatacept arm is smaller than or equal to 12%. Estimate and 95% confidence interval (CI) for difference based on minimum risk weights method with randomization stratification of screening Disease Activity Score-28 (DAS28) c-reactive protein (CRP); minimum risk weights method; adjusted for randomization stratification of screening Disease Activity Score-28 (DAS28) c-reactive protein (CRP); Difference from adalimumab at Day 365 = 1.8, 95% CI 2-sided [-5.6 to 9.2]

2. Secondary Outcome: Proportion of Participants With Local Injection Site Reactions Adverse Events (Pre-specified) Reported During 12 Month Period - ITT Population
Description: n=number of participants with a pre-specified local injection site reaction event, N=number of participants at risk. Proportion (%) = n/N. 12 Months includes data up to 56 days post last dose of the first 12 months Period or start of the first dose of second 12 months period.
Time Frame: Day 1 to 12 Months
Population: The ITT analysis population was defined as all participants randomized into the study who received at least one dose of study drug. n/N = 12/318, 30/328 in abatacept and adalimumab, respectively. CI based on normal approximation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abatacept | Adalimumab
Number analyzed (Participants) | 318 | 328
percentage of participants | 3.8 [1.68 to 5.87] | 9.1 [6.03 to 12.27]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab; Analysis is p-value of difference in proportions. n=number of participants with event, N=number of participants at risk. Proportion = n/N. In order to maintain the overall type I error rate of 0.05 for testing both the primary non-inferiority hypothesis and the key secondary local injection site reaction (LISR) hypothesis, the LISR hypothesis was tested at the 5% significance level only after the primary non-inferiority hypothesis is established at the 5% level; Test type: Superiority or Other; p = 0.006, Chi-squared; Difference in proportions = -5.37, 95% CI 2-sided [-9.13 to -1.62]

3. Secondary Outcome: Incidence Rate of Local Injection Site Reactions (Pre-specified) Reported During 24 Month Period - ITT Population
Description: Incidence Rate: (incidence/100 person-years) = number of participants with event * 100 /exposure (person-years) Exposure (person-years) = the sum over all participants of the exposure per participant in the 24 months (censored at the time of first occurrence of AE) expressed in days, divided by 365.25. The 24 Month Period includes data up to 56 days post the last dose in the 24 month period. Poisson distribution used to construct the 95% CIs.
Time Frame: Day 1 to Day 729
Population: ITT population: all participants randomized into the study who received at least one dose of study drug. Participants with a pre-specified local injection site event at 24 Months: 13, 34, in abatacept and adalimumab arms, respectively. 24 Month Exposure=579.21, 532.99, respectively.
Measure: Number (95% Confidence Interval); unit: incidence/100 person years
Arm/Group | Abatacept | Adalimumab
Number analyzed (Participants) | 318 | 328
incidence/100 person years | 2.24 [1.20 to 3.84] | 6.38 [4.42 to 8.91]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab; Analysis of incidence rate at 24 months. Point estimate and 95% CI. Poisson distribution was used to construct the 95% CIs; Test type: Superiority or Other; Difference from adalimumab = -4.13, 95% CI 2-sided [-6.55 to -1.72]

4. Secondary Outcome: Proportion of Participants Without Radiographic Progression in Total Score Less Than or Equal to the Smallest Detectable Change (SDC) From Baseline to Months 12 and 24 Using Modified Van Der Heijde Total Sharp Score (mSvdHS) - ITT Population
Description: Plain radiographs of hands and feet taken at baseline (BL), Day 365, and Day 729. BL and Day 365 radiographs were re-read concurrent with Day 729 films by readers blinded to sequence and treatment (a second pre-specified reading campaign). SDC defined as amount of change for which anything smaller could not be reliably distinguished from random error in measurement of simultaneously read films. Non-progression defined: change from BL (Day 1, prior to dosing) in total score less than, equal to (<=) SDC(2.2). Proportion n/m (%)=number meeting criteria (n); number analyzed (m). SDC calculated as SD/sqrt(2)*1.96/sqrt(2)with standard deviation (SD) of paired differences of change from BL in total score between 2 readers; squared root(sqrt). mSvdHS=summary of erosion severity in 32 hand and 12 foot joints. Hand joints scored 0 to 5; foot joints 0 to 10 with 0=no erosion and higher numbers indicating greater erosion severity. BL: radiographic data within 14 days or less of first dose.
Time Frame: Baseline to Day 729
Population: ITT population: all subjects randomized into the study who received at least one dose of study drug. Number analyzed: m=number of ITT participants with both BL and post-BL total score: Day 365: m=295, 297;Day 729 m=257 and 260, in abatacept and adalimumab arms, respectively. n=number without progression. CI based on normal approximation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abatacept | Adalimumab
Number analyzed (Participants) | 295 | 297
percentage of participants
  Day 365 n=259, 263; m=295, 297 | 87.8 [84.1 to 91.5] | 88.6 [84.9 to 92.2]
  Day 729 n=218, 218; m=257, 260 | 84.8 [80.4 to 89.2] | 83.8 [79.4 to 88.3]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab; This analysis is for Day 365; Test type: Superiority or Other; minimum risk weights method; Adjusted for randomization stratification of screening Disease Activity Score-28 (DAS28) c-reactive protein (CRP); Difference from adalimumab at Day 365 = -1.3, 95% CI 2-sided [-6.5 to 3.9]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab; This analysis is for Day 729; Test type: Superiority or Other; minimum risk weights method; Adjusted for randomization stratification of screening Disease Activity Score-28 (DAS28) c-reactive protein (CRP); Difference from adalimumab at Day 729 = 0.9, 95% CI 2-sided [-5.5 to 7.3]

5. Secondary Outcome: Incidence Rate of Serious Adverse Events (SAEs), Serious Infections, Pre-specified Opportunistic Infections, and Discontinuation for Any Cause at 12 Months of Treatment - ITT Population
Description: Pre-specified opportunistic infections include: pneumonia, tuberculosis, herpes zoster, combined opportunistic infections, all hospitalized infections. Incidence Rate: incidence/100 person-years: numerator was number of unique events within this period (up to 56 days post-last dose of first 12 months or start of first dose of second 12 months); denominator was overall total exposure (person-years) within this period, calculated as sum over all participants of exposure (in days) divided by 365.25. The resulting incidence rate was multiplied by 100 to express rate per 100 person-years. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE is a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: Day 1 to Day 365
Population: The intent to treat (ITT) analysis population was defined as all subjects randomized into the study who received at least one dose of study drug. Poisson distribution was used to construct the 95% CIs.
Measure: Number (95% Confidence Interval); unit: incidence/100 person-years
Arm/Group | Abatacept | Adalimumab
Number analyzed (Participants) | 318 | 328
incidence/100 person-years
  SAE (number with event=32, 30) | 11.06 [7.57 to 15.62] | 10.26 [6.92 to 14.65]
  Serious Infections (number with event=7, 9) | 2.32 [0.93 to 4.79] | 2.99 [1.37 to 5.68]
  Opportunistic infections (number with event=1, 1) | 0.33 [0.01 to 1.83] | 0.33 [0.01 to 1.85]
  Discontinuation (number with event=44, 59) | 14.79 [10.74 to 19.85] | 20.11 [15.31 to 25.94]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab; Analysis for incidence rate of SAE at 12 months. Point estimate and 95% CI for treatment difference. Poisson distribution was used to construct the 95% CIs; Test type: Superiority or Other; Difference from adalimumab = 0.80, 95% CI 2-sided [-4.51 to 6.11]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab; Analysis for incidence rate of Serious Infections and Infestations at 12 months. Point estimate and 95% CI for treatment difference. Poisson distribution was used to construct the 95% CIs; Test type: Superiority or Other; Difference from adalimumab = -0.67, 95% CI 2-sided [-3.27 to 1.94]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab; Analysis for incidence rate of Opportunistic Infections at 12 months. Point estimate and 95% CI for treatment difference. Poisson distribution was used to construct the 95% CIs; Test type: Superiority or Other; Difference from adalimumab = -0.00, 95% CI 2-sided [-0.92 to 0.91]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab; Analysis for incidence rate of discontinuation for any cause at 12 months. Point estimate and 95% CI for treatment difference. Poisson distribution was used to construct the 95% CIs; Test type: Superiority or Other; Difference from adalimumab = -5.32, 95% CI 2-sided [-12.06 to 1.41]

6. Secondary Outcome: Incidence Rate of Serious Adverse Events (SAEs), Serious Infections, Pre-specified Opportunistic Infections, and Discontinuation for Any Cause at 24 Months of Treatment - ITT Population
Description: Pre-specified opportunistic infections include: pneumonia, tuberculosis, herpes zoster, combined opportunistic infections, and all hospitalized infections. Incidence Rate: incidence/100 person-years: numerator was number of unique events within this period (up to 56 days post the last dose of the 24 Months period); denominator was overall total exposure (person-years) within this period, which was calculated as the sum over all participants of exposure (in days) divided by 365.25. The resulting incidence rate was multiplied by 100 to express the rate per 100 person-years. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE is a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: Day 1 to Day 729
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: incidence/100 person-years
Arm/Group | Abatacept | Adalimumab
Number analyzed (Participants) | 318 | 328
incidence/100 person-years
  SAE Incidence Rate (number with event=44, 54) | 13.8 [10.04 to 17.63] | 16.5 [12.45 to 20.48]
  Serious Infections (number with event=12, 19) | 3.8 [1.68 to 5.87] | 5.8 [3.26 to 8.32]
  Opportunistic infections (number with event=2, 5) | 0.6 [0.00 to 1.50] | 1.5 [0.20 to 2.85]
  Discontinuation (number with event=66, 83) | 20.8 [16.30 to 25.21] | 25.3 [20.60 to 30.01]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab; Analysis for incidence rate of SAE at 24 months. Point estimate and 95% CI for treatment difference. Poisson distribution was used to construct the 95% CIs; Test type: Superiority or Other; Difference from adalimumab = -1.91, 95% CI 2-sided [-5.43 to 1.61]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab; Analysis for incidence rate of Serious infections and infestations Adverse Events at 24 months. Point estimate and 95% CI for treatment difference. Poisson distribution was used to construct the 95% CIs; Test type: Superiority or Other; Difference from adalimumab = -1.24, 95% CI 2-sided [-3.12 to 0.63]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab; Analysis for incidence rate of opportunistic infections at 24 months. Point estimate and 95% CI for treatment difference. Poisson distribution was used to construct the 95% CIs; Test type: Superiority or Other; minimum risk weights method; Difference from adalimumab = -0.52, 95% CI 2-sided [-1.39 to 0.36]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab; Analysis for incidence rate of discontinuations (all cause) at 24 months. Point estimate and 95% CI for treatment difference. Poisson distribution was used to construct the 95% CIs; Test type: Superiority or Other; Difference from adalimumab = -3.10, 95% CI 2-sided [-7.13 to 0.92]

7. Secondary Outcome: Proportion of Participants With Induction of Autoantibodies During the 12 Months and 24 Months Periods - ITT Population
Description: The induction of autoantibodies was defined as participant's antinuclear antibodies (ANA) or anti-double stranded deoxyribonucleic acid (dsDNA) converting from a negative status at baseline to a positive status at a post-baseline measurement time point (Day 365 or Day 729). Proportion (%) = n/m, where n=number of participants with positive ANA or dsDNA at a time point and m=number of participants who had negative ANA or dsDNA at baseline. Blood samples were first tested for ANA by indirect fluorescent assay using HEp-2 Cell Line Substrate, and when positive, samples were further tested for anti-dsDNA by indirect fluorescent assay using Crithidia Luciliae Substrate.
Time Frame: Day 1 to Day 729
Population: ITT population was defined as all participants randomized into the study who received at least one dose of study drug; number analyzed was ITT participants with data at each time point and who had negative ANA or dsDNA at baseline (m)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Adalimumab
Number analyzed (Participants) | 318 | 328
Percentage of participants
  Day 365 ANA; n=12, 28; m=229, 210 | 5.2 [2.4 to 8.1] | 13.3 [8.7 to 17.9]
  Day 365 anti-dsDNA; n=1, 29; m=299, 293 | 0.3 [0.0 to 1.0] | 9.9 [6.5 to 13.3]
  Day 729 ANA; n=12, 24; m=190, 163 | 6.3 [2.9 to 9.8] | 14.7 [9.3 to 20.2]
  Day 729 anti-dsDNA; n=0, 29; m=248, 237 | 0.0 [0.0 to 0.0] | 12.2 [8.1 to 16.4]
Statistical Analysis 1: Comparison: Abatacept vs Adalimumab; Analysis for ANA at Day 365. Point estimate and 95% CI for treatment difference; Test type: Superiority or Other; Difference from adalimumab = -8.1, 95% CI 2-sided [-13.9 to -2.2]
Statistical Analysis 2: Comparison: Abatacept vs Adalimumab; Analysis for ANA at Day 729. Point estimate and 95% CI for treatment difference; Test type: Superiority or Other; Difference from adalimumab = -8.4, 95% CI 2-sided [-15.3 to -1.5]
Statistical Analysis 3: Comparison: Abatacept vs Adalimumab; Analysis for dsDNA at Day 365. Point estimate and 95% CI for treatment difference; Test type: Superiority or Other; Difference from adalimumab = -9.6, 95% CI 2-sided [-13.4 to -5.7]
Statistical Analysis 4: Comparison: Abatacept vs Adalimumab; Analysis for dsDNA at Day 729. Point estimate and 95% CI for treatment difference; Test type: Superiority or Other; Difference from adalimumab = -12.2, 95% CI 2-sided [-16.9 to -7.6]

ADVERSE EVENTS:
Time Frame: Includes data up to 56 days post the last dose in the 24 months period.
Description: Note: One participant in the abatacept arm had an SAE with no preferred term identified. Therefore, there were 44 participants with SAEs reported in the Outcome measure on the Rate of SAEs but since a preferred term was not identified, a total of 43 are identified in the SAEs below.
Arm/Group | Abatacept | Adalimumab
Serious Adverse Events (participants affected / at risk) | 43/318 | 54/328
Other Adverse Events (participants affected / at risk) | 237/318 | 232/328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept (N=318) | Adalimumab (N=328)
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Drug dependence (Psychiatric disorders) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0
Hernia obstructive (General disorders) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 2
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Groin abscess (Infections and infestations) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 3
Palpitations (Cardiac disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Convulsion (Nervous system disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 3 | 0
Clostridial infection (Infections and infestations) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Human papilloma virus test positive (Investigations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 4
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis bacterial (Infections and infestations) | 0 | 3
Bursitis infective staphylococcal (Infections and infestations) | 0 | 1
Chest pain (General disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Disseminated tuberculosis (Infections and infestations) | 0 | 1
Histoplasmosis disseminated (Infections and infestations) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Chest wall abscess (Infections and infestations) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Angina pectoris (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept (N=318) | Adalimumab (N=328)
Fatigue (General disorders) | 21 | 20
Headache (Nervous system disorders) | 32 | 38
Diarrhoea (Gastrointestinal disorders) | 29 | 23
Gastroenteritis (Infections and infestations) | 16 | 13
Nasopharyngitis (Infections and infestations) | 61 | 57
Sinusitis (Infections and infestations) | 51 | 37
Vomiting (Gastrointestinal disorders) | 11 | 18
Rash (Skin and subcutaneous tissue disorders) | 13 | 27
Upper respiratory tract infection (Infections and infestations) | 64 | 55
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 39
Nausea (Gastrointestinal disorders) | 26 | 28
Influenza (Infections and infestations) | 21 | 18
Oedema peripheral (General disorders) | 22 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 17
Bronchitis (Infections and infestations) | 49 | 43
Depression (Psychiatric disorders) | 17 | 14
Pharyngitis (Infections and infestations) | 17 | 20
Urinary tract infection (Infections and infestations) | 41 | 32
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 27
Hypertension (Vascular disorders) | 21 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.